CLINICAL TRIAL: NCT02158286
Title: Validation of Paracetamol Absorption Technique as a Method for Measuring Gastric Tube Outlet to Golden Standard, to Scintigraphy. A Pilot Study
Brief Title: Paracetamol Absorption Technique as a Method for Measuring Gastric Tube Outlet
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: TS2010
Record Dates: First submitted 2014-06-02; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Esophageal and/or Cardia Cancer; Esophagectomy; Gastric Pull-up Reconstruction

STUDY DESIGN:
Observational Model: Case-Only

GROUPS / COHORTS (1):
- Esophagectomy, Emptying from gastric tube: Validate paracetamol clearance technique to scintigraphy for measuring emptying rate from the gastric tube.
  Interventions: Other: Measuring emptying rate from the gastric tube

INTERVENTIONS:
Other: Measuring emptying rate from the gastric tube
  Other Names: Paracetamol clearance technique; Scintigraphy

SUMMARY:
Retention of the gastric tube after esophagectomy is a clinically important problem, and there is a need of a simple method to evaluate emptying rate from the gastric tube after esophagectomy. Scintigraphy is the golden standard of measuring emptying rate from the gastric tube. In non-operated patients, paracetamol clearance technique have been widely used for measuring gastric emptying rate. There is no validation however if paracetamol clearance technique can be used for measuring emptying rate of the gastric tube. The investigators aim of this pilot- study is to validate paracetamol clearance technique to scintigraphy for measuring emptying rate from the gastric tube and to evaluate if there is a correlation between symptoms of retention and quality of life with the emptying rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients where it had past at least two years since they had underwent an Ivor Lewis esophagectomy with gastric pull-up reconstruction.
* no signs of recurrence
* >18 years of age

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients where it had past at least two years since they had underwent an Ivor Lewis esophagectomy with gastric pull-up reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Validate paracetamol clearance technique to scintigraphy for measuring emptying rate from the gastric tube | Up to 12 months
  During one diagnostic measurement perform, simultaneously, scintigraphy and paracetamol clearance technique to measure emptying rate from the gastric tube. After the test the patient answer both a QOL questionnaire and symptom questionnaire.

SECONDARY OUTCOMES:
Evaluate if patient with symptoms of slow emptying rate from the gastric tube also have slow emptying rate measured with scintigraphy. | Up to 12 months
  Patients will answer the questionaire EORTC QLQ OG25 for validation of upper gastrointestinal symptoms and the questionnaire EORTC QLQ C30 for validation of quality of life. Emptying rate from the gastric tube is measured with scintigraphy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Lund, Sweden